CLINICAL TRIAL: NCT04433364
Title: COPE - COVID-19 in Pregnancy and Early Childhood - a Study Protocol for a Prospective Multicentre Cohort Study
Brief Title: COPE - COVID-19 in Pregnancy and Early Childhood
Acronym: COPE
Status: Active, not recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Verena Sengpiel, MD, PhD, Senior Consultant, Sahlgrenska University Hospital
Other Study IDs: 2020-02848 0604
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Sars-CoV2; Covid-19; Pregnancy Complications; Pregnancy Preterm; Pregnancy in Diabetic; Neonatal Infection
Keywords: sars-cov2; covid-19; pregnancy; neonatal; long-term follow-up; complications
MeSH Terms: conditions — COVID-19; Pregnancy Complications; Pregnancy in Diabetics | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples Without DNA — Bloodsample from the mother antenatally, at inclusion and at delivery from healthy women, as well as NPH-swab and placenta at delivery. Naval cord blood from healthy infants. From covid-19 pos women: blood sample antenatally and at diagnosis as well as vaginal, rectal and NPH swab and urinary sample. At delivery NPH-swabs as well as vaginal and rectal swabs and urinary samples and blood and in case of caesarean section amnion fluid and spinal fluid. Breastmilk at 48-96 hours after delivery. From the infant naval cord blood and at 48-96 hours after delivery NPH-swab and rectal swab as well as blood sample. For the COVID-19 group a follow-up visit during the first year after delivery for bloodsamples of mother and child/children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screening group: a general population of women giving birth, called "screening group" included at routine antenatal visits, their partners, and children
  Interventions: Other: biological samples, questionnaires and interviews
- COVID-19 group: group of women testing positive for SARS-CoV-2 or falling ill with COVID-19, called "COVID-19 group", their partners, and children
  Interventions: Other: biological samples, questionnaires and interviews

INTERVENTIONS:
Other: biological samples, questionnaires and interviews — Biological samples: to study impact of testing positive for SARS-CoV-2 during pregnancy samples taken in routine clinical care, samples from already existing research biobanks and the newly established COPE biobank will be used. Time-points: inclusion, at delivery mother and fetus. Covid-19 positive group only: 48-96 h, 2 months postpartum for mother and fetus.
  Questionnaires: Women and partners in both groups will fill out electronical questionnaires at different time points during pregnancy and until 12 months postpartum based on validated instruments to test for differences in Self-Efficacy, Anxiety and Depression, Health-related quality of life, Sense of Coherence, PTSD Symptoms, Postpartum Bonding, Childbirth experiences and Self-Efficacy of Breastfeeding. The child's health will be assessed regarding infection until 6 weeks of age and development until 4 years.
  Interviews: 24-40 women and partners in both groups. Interviews will be conducted 3 to 6 months after childbirth.

SUMMARY:
Purpose: The emergence of a new coronavirus SARS-CoV-2 causing a novel infection in the human race resulting in a world-spanning pandemic came as a surprise and at a tremendous cost both for individual human lives as well as for the society and the health care sector. The knowledge on how this new infection affects both the mother and the unborn child as well as the outcomes for the mother and the child in the long run are unknown. What is known is based on case-reports and small case-series solely. Both the coronaviruses causing Middle East Respiratory Syndrome (MERS) and Severe Acute Respiratory Syndrome (SARS) can cause a threat to pregnant women and their offspring, which leads to the question whether this could be the case also for SARS-CoV-2.

Aims: To establish a biobank of biological material from infected as well as non-infected pregnant women and their offspring. To combine this biobank with Swedish quality and health care registers, computerized patient charts and questionnaire data, enabling both short-term follow up, such as obstetric outcomes, as well as long-term outcomes both for mother and child. To study how the pandemic situation affects both the mother and her partner in their experience of pregnancy, childbirth, and early parenthood.

Design: A national Swedish multicentre study. Women are included when they have a positive test for SARS-CoV-2 or a clinical suspicion of coronavirus disease 2019 (COVID-19) (COVID-19 group). Pregnant women without COVID-19 symptoms will be included at their routine visits (Screening group). Blood samples and other biological material will be collected at different time-points. Additional predictors and outcomes are collected from the Swedish Pregnancy Register as well as obligatory Swedish health registers. The biobank and its linkage to health registers through the Swedish personal identification number will enable future research. Child development will be followed during the first year of life by questionnaires to the parents. Womens' and their partners' experience of childbirth and parenthood will be studied in form of questionnaires as well as in form of interviews.

Conclusion: This project will help obstetricians and neonatologists better recognize clinical manifestations of the virus, identify possible risk factors during pregnancy and tailor therapies alongside providing right level of surveillance and management during pregnancy, delivery, and child health care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years of age and above
* Attending routine antenatal visits at a participating hospital during the study period or are strongly suspicious of or diagnosed with Covid-19 during pregnancy.
* For the questionnaire part: language knowledge (Swedish, English, Arabic, Somali)
* For the interview part: Swedish language knowledge

Exclusion Criteria:

• Another language but selected ones

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 years of age and above. Attending routine antenatal visits at a participating hospital during the study period or are strongly suspicious of or diagnosed with Covid-19 during pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 3834 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Biobank with linkage to registers | 1-20 years
  establish a biobank and database with bio-samples from both women that are not tested and presumed healthy as well as possibly ill and women confirmed tested positive for SARS-CoV-2 and their infants linked to Swedish health care registers including socio-economic factors and use serological and viral analyses from the biological samples to evaluate maternal, fetal and neonatal outcomes.
Experiences of pregnancy during a pandemic | 1 year
  study how women and their partners experience pregnancy, childbirth and early parenthood in the COVID-19-pandemic, both for women not tested and for women tested positive for SARS-CoV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Verena Sengpiel, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (27):
- Sweden (27):
  - Falu Hospital, Falun, Dalarna County
  - Halmstad lasarett, Halmstad, Halland County
  - Varbergs sjukhus, Varberg, Halland County
  - Helsingborgs lasarett, Helsingborg, Skåne County
  - Skåne Universitetssjukhus, Lund, Skåne County
  - Eskiltuna hospital, Eskilstuna, Södermanland County
  - Boras hospital, Borås, VGR
  - Sahlgrenska Univeristy Hospital, Gothenburg, VGR
  - Ryhovs sjukhus, Jönköping
  - Kalmar Lasarett, Kalmar
  - Karlstad lasarett, Karlstad
  - Kristiandstad länssjukhus, Kristianstad
  - Örebro University Hospital, Örebro
  - Skaraborgs sjukhus Skövde, Skövde
  - BB Stockholm, Stockholm
  - Danderyd, Stockholm
  - Karolinska University Hospital Solna, Stockholm
  - Karolinska University Hospital- Huddinge, Stockholm
  - Södersjukhuset, Stockholm
  - Södertälje, Stockholm
  - Sundsvall, Sundsvall
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Västerås, Västerås
  - Ystad, Ystad
  - Linköping University Hospital, Linköping, Östergötland County
  - Vrinnevisjukhuset, Norrköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Yes
Outcome variables
Supporting Information: Study Protocol, ICF
Time Frame: 2024
Access Criteria: Ethical permission
URL: http://www.copestudien.se

REFERENCES:
- [Derived] Carlsson Y, Bergman L, Zaigham M, Linden K, Andersson O, Veje M, Sandstrom A, Wikstrom AK, Ostling H, Fadl H, Domellof M, Blomberg M, Brismar Wendel S, Aden U, Sengpiel V; COPE study group. COVID-19 in Pregnancy and Early Childhood (COPE): study protocol for a prospective, multicentre biobank, survey and database cohort study. BMJ Open. 2021 Sep 14;11(9):e049376. doi: 10.1136/bmjopen-2021-049376. PMID 34521667